CLINICAL TRIAL: NCT03843047
Title: Effects of Electronic Cigarette Unit Price Manipulations in the Experimental Tobacco Marketplace on Tobacco Product Substitution
Brief Title: Electronic Cigarette Unit Price Manipulations in the Experimental Tobacco Marketplace
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Principal Investigator, Jeffrey Stein, Research Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 18-268
Record Dates: First submitted 2019-02-12; First posted 2019-02-15 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Tobacco Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Intervention Model Description: Participants will complete different purchasing scenarios in the Experimental Tobacco Marketplace in which different e-liquid nicotine concentrations are available (3, 6, 12, and 24 mg/mL nicotine). In all scenarios, a range of other tobacco products will also be available.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dual cigarette smokers/e-cigarette users (Other): Dual cigarette smokers/e-cigarette users will be recruited.
  Interventions: Drug: 3 mg/mL nicotine strength e-liquid; Drug: 6 mg/mL nicotine strength e-liquid; Drug: 12 mg/mL nicotine strength e-liquid; Drug: 24 mg/mL nicotine strength e-liquid
- Exclusive cigarette smokers (Other): Exclusive cigarette smokers with minimal prior e-cigarette experience will be recruited.
  Interventions: Drug: 3 mg/mL nicotine strength e-liquid; Drug: 6 mg/mL nicotine strength e-liquid; Drug: 12 mg/mL nicotine strength e-liquid; Drug: 24 mg/mL nicotine strength e-liquid

INTERVENTIONS:
Drug: 3 mg/mL nicotine strength e-liquid — Availability of 3 mg/mL nicotine strength e-liquid in the Experimental Tobacco Marketplace
Drug: 6 mg/mL nicotine strength e-liquid — Availability of 6 mg/mL nicotine strength e-liquid in the Experimental Tobacco Marketplace
Drug: 12 mg/mL nicotine strength e-liquid — Availability of 12 mg/mL nicotine strength e-liquid in the Experimental Tobacco Marketplace
Drug: 24 mg/mL nicotine strength e-liquid — Availability of 24 mg/mL nicotine strength e-liquid in the Experimental Tobacco Marketplace

SUMMARY:
Electronic cigarettes (e-cigarettes) may be a safer alternative to conventional cigarettes and are available in a broad range of nicotine strengths. The overall goal of this project is to use an experimental analogue of the real-world tobacco marketplace to examine the effects of nicotine strength on e-cigarette consumption and the likelihood that current smokers will either switch to e-cigarettes (which may reduce harm) or use both products in combination (which may increase harm). Testing effects of e-cigarette nicotine strength under controlled conditions in a context that models the real world will facilitate evidence-based policies that have a net benefit to health.

DETAILED DESCRIPTION:
The goal of tobacco regulation is to reduce tobacco-related harm and improve public health. Improving public health in this way requires thorough understanding of the processes underlying purchasing and consumption of the various products available in the complex tobacco marketplace. One product feature eligible for regulation is the nicotine content in electronic cigarettes (e-cigarettes). At present, little research has experimentally examined the influence of nicotine strength on e-cigarette consumption and the likelihood that current cigarette smokers will switch to e-cigarettes (i.e., product substitution). In the absence of such evidence, regulation designed to restrict available e-cigarette nicotine strength may have unanticipated consequences. This project will utilize an innovative method, the Experimental Tobacco Marketplace, to provide estimates of the effects of e-cigarette nicotine strength on tobacco consumption and the degree to which e-cigarette products serve as functional substitutes for cigarettes. In so doing, this project will provide rigorous tests of a novel quantitative model able to account for e-cigarette substitution effects, including effects of nicotine strength. This model, which assumes that product substitution is directly influenced by the nicotine content of tobacco products relative to their prices (a phenomenon called unit price), provides a framework that may be used to generate novel predictions and guide regulatory efforts. This project will examine the effects of four e-cigarette nicotine strengths (3, 6, 12, and 24 mg/mL) on the degree to which e-liquid substitutes for conventional cigarettes in the Experimental Tobacco Marketplace. This project will examine these effects in: a) exclusive cigarette smokers with minimal prior e-cigarette experience, and b) dual cigarette smokers/e-cigarette users. Together, the findings from this project may be used to inform regulatory action and will improve understanding of the role of nicotine strength in determining the extent to which e-cigarettes serve as functional substitutes for conventional cigarettes.

ELIGIBILITY:
Inclusion Criteria:

* Current cigarette smoker
* Current e-cigarette user (dual users arm) or have minimal prior e-cigarette experience (exclusive smokers arm)
* Cotinine levels that confirm tobacco use
* Willing to try e-cigarettes

Exclusion Criteria:

* Unstable psychiatric or medical conditions
* Immediate plans to quit smoking
* Use of prescription medication that might affect smoking or nicotine metabolism
* Pregnancy (females)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
E-liquid substitution | 1 day
  The degree to which various e-liquid nicotine strengths (3, 6, 12, 24 mg/mL) substitute for conventional cigarettes will be assessed.

SECONDARY OUTCOMES:
Cigarette demand | 1 day
  The degree to which various e-liquid nicotine strengths (3, 6, 12, 24 mg/mL) influence demand form conventional cigarettes will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Jeff S. Stein, Ph.D., Principal Investigator — Fralin Biomedical Research Institute at VTC
Locations (1):
- Fralin Biomedical Research Institute, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided